CLINICAL TRIAL: NCT06665360
Title: Sound Timbre-based Milling Status Identification in Robotic Vertebral Lamina Milling
Brief Title: Identify the State of Laminae Milling by Sound
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Nankai University (Other)
Responsible Party: Principal Investigator, Rui Wang, Ph.D. Candidate, Tianjin Medical University General Hospital
Other Study IDs: IRB2021-KY-198
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Spinal Degenerative Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- posterior spinal decompression
  Interventions: Other: The high speed bur was used to mill the cancellous cortical bone of the lamina

INTERVENTIONS:
Other: The high speed bur was used to mill the cancellous cortical bone of the lamina — The high speed bur was used to mill the cancellous cortical bone of the lamina

SUMMARY:
After verifying the signals collected in the laboratory, the investigators performed a preliminary verification in the surgery, in which the sound pressure signals of lamina milling were collected during the surgery to identify milling status.

DETAILED DESCRIPTION:
The sound of milling cortical bone and cancellous bone were recorded during posterior spinal decompression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with myelopathy caused by spinal stenosis who had undergone posterior decompression.

Exclusion Criteria:

1. Receipt of surgery using an anterior approach or circumferential spinal cord decompression through a posterior approach;
2. Experience of trauma;
3. History of spinal tumor;
4. Previous spinal surgery;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with spinal stenosis requiring surgery
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Amplitude of sound pressure | The sound pressure signals were collected during the operation in 6 cases, an average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided